CLINICAL TRIAL: NCT07196163
Title: An Exploratory Clinical Study of Golidocitinib in Adult Patients With Primary Immune Thrombocytopenia (ITP)
Brief Title: An Exploratory Study of Golidocitinib in Adult Patients With ITP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Associate Director, Peking University People's Hospital
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DZ2024J0003
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: Part A-Open-label Sequential, Part B-Double-blind Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A-Open-label, Part B-Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Golidocitinib Part B (Experimental): Golidocitinib at recommended phase 2 doses, administered orally, once daily.
  Interventions: Drug: Golidocitinib
- Placebo Part B (Placebo Comparator): Placebo at recommended phase 2 doses, administered orally, once daily.
  Interventions: Drug: Placebo
- Golidocitinib Part A (Experimental): Golidocitinib dose escalation, administered orally, once daily.
  Interventions: Drug: Golidocitinib

INTERVENTIONS:
Drug: Golidocitinib — Golidocitinib will be administered orally as capsules in a 28-day cycle.
  Arms: Golidocitinib Part A; Golidocitinib Part B
Drug: Placebo — Placebo will be administered orally as capsules in a 28-day cycle.
  Arms: Placebo Part B

SUMMARY:
This is a multicenter clinical study to evaluate the safety and efficacy of golidocitinib in patients with primary immune thrombocytopenia (ITP). The study consists of two parts: Part A dose escalation and Part B dose expansion. Part A is designed to obtain the safety profile of golidocitinib in patients with ITP and the recommended dose for the randomized cohort in Part B. Part B is a randomized, double-blind, placebo-controlled study, and the primary objective of this part is to evaluate the preliminary efficacy of golidocitinib in patients with ITP.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 18 and 80 years old.
* Primary ITP for >3 months.
* An average of two platelet counts (⩾ 7 days apart) of < 30 × 10⁹/L.
* Have relapsed or treatment-resistant to previous ITP therapies, including corticosteroids and at least one other ITP therapy.
* Have history of response to previous treatments.
* Adequate hematologic, hepatic, and renal fuction.
* Participants willing to comply with contraceptive restrictions.

Exclusion Criteria:

* Diagnosed with secondary immune thrombocytopenia, or there is evidence that the patient has a secondary cause of immune thrombocytopenia.
* Previous or current therapy and comedications meet exclusion criteria.
* Patients with major caridiovascular disease, active infetion, maligancy or uncontrolled systemic disease.
* Women who are breast feeding.
* History of hypersensitivity to sudy drug with a similar chemical structure or class.
* Previously received JAK inhibitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence and severity of Adverse Events (AEs) | 1 year
  The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events.
Part B: Durable response rate | up to 24 weeks
  The proportion of patients with a platelet count ≥ 50 × 10⁹/L on at least four of six scheduled visits between weeks 14 and 24

SECONDARY OUTCOMES:
Part A: Durable response rate | up to 24 weeks
  The proportion of patients with a platelet count ≥ 50 × 10⁹/L on at least four of six scheduled visits between weeks 14 and 24
Part B: Incidence and severity of Adverse Events (AEs) | 1 year
  The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events.
Part A and Part B: Overall response rate | up to 24 weeks
  The proportion of patients with a platelet count ≥ 100 × 10⁹/L on 2 consecutive visits at least 7 days apart and without bleeding
Part A and Part B: Complete response rate | up to 24 weeks
  The proportion of patients with a platelet count ≥ 100 × 10⁹/L on 2 consecutive visits at least 7 days apart and without bleeding
Part A and Part B: Early response rate | up to 1 week
  The proportion of patients with a platelet count ≥ 30 × 10⁹/L and doubling of the baseline count and without bleeding within 1 week
Part A and Part B: Initial response rate | up to 4 weeks
  The proportion of patients with a platelet count ≥ 30 × 10⁹/L and doubling of the baseline count and without bleeding within 4 weeks
Part A and Part B: Sustained response rate | up to 24 weeks
  The proportion of patients with a platelet count ≥ 30 × 10⁹/L and doubling of the baseline count and without bleeding between weeks 20 and 24
Part A and Part B: Time to response | up to 24 weeks
  Time to first platelet counts ≥ 30 × 10⁹/L and doubling of the baseline count and without bleeding
Part A and Part B: Cumulative response time | up to 24 weeks
  Number of cumulative days with platelet counts ≥ 30 × 10⁹/L and doubling of the baseline count and without bleeding by Week 24
Part A and Part B: The proportion of patients requiring rescue therapy | up to 24 weeks
Part A and Part B: The proportion of patients experencing bleeding (≥ Grade 2) | up to 24 weeks
Part A and Part B: Changes of ITP-BAT bleeding score | up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No